CLINICAL TRIAL: NCT05041868
Title: Physical Rehabilitation in Women With Scleroderma: Effects on Pulmonary Function, Lung Ultrasound, Muscle Function, Hand Functional, Functional Capacity, and Quality of Life
Brief Title: Rehabilitation Program in Patients With Scleroderma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitário Augusto Motta (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 02794918.1.0000.5259
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-07

CONDITIONS: Scleroderma; System; Sclerosis; Muscle Strain; Physical Disability; Quality of Life; Exercise
Keywords: Scleroderma; Physical Therapy; Rehabilitation; Functional capacity; Exercise; ADL-Glittre test
MeSH Terms: conditions — Scleroderma, Diffuse; Sprains and Strains; Motor Activity | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Women with Scleroderma will use a booklet-guided rehabilitation program that lasts three months (3 times per week with a duration of 60 minutes per session). Consisting of stretching, warm-up and cool-down exercises, muscle strengthening (flexion, extension, adduction, and abduction movements in exercises involving open and closed kinetic chains), endurance exercises, aerobic training, balance training and proprioception. The patient will be evaluated at 2 different timepoints (baseline and after 12 weeks of training). The physiotherapist contacts the patient by phone weekly to follow the progression of the treatment. Before and after the intervention, patients will be submitted to the following assessments: Cochin Hand Functional Scale (CHFS), Short-Form 36 Health Survey (SF-36); Scleroderma Health Assessment Questionnaire Disability Index (SHAQ-DI); lung function; lung ultrasound; handgrip; Glittre Activities of Daily Living test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): The program comprises the practice of warm-up, muscle strengthening with free weights and with their own body weight against the action of gravity for the main muscular groups, balance control training, aerobic training, and relaxation exercises. The proposal consists of 3 weekly sessions, for 12 consecutive weeks.
  Interventions: Other: Treatment

INTERVENTIONS:
Other: Treatment — After a physical therapy evaluation, the patient underwent a booklet-guided physical exercise program that lasted three months (3 times per week with a duration of 60 minutes per session). Activities included overall stretching and strengthening (flexion, extension, adduction and abduction movements) and muscular endurance exercises (exercises involving open and closed kinetic chains), along with aerobic conditioning using a functional circuit. The patient was evaluated at 2 different timepoints (baseline and after treatment). The physiotherapist contacted the patient by phone weekly to follow the progression of the treatment.

SUMMARY:
Scleroderma (or Systemic Sclerosis - SSc) is one of the most neglected diseases worldwide, according to the World Health Organization. In the adult population with SS, the systemic effects of the disease, such as respiratory and peripheral muscle dysfunction, cause a decrease in quality of life. As a consequence, there is a concern about functional rehabilitation, since the aging of this population is already a reality. Thus, the objective of this project is to evaluate the effects of functional rehabilitation on functional capacity and quality of life in women over 18 years of SS. In this longitudinal intervention study, patients will be submitted to a three-month rehabilitation program. Before and after the intervention, patients will be submitted to the following assessments: Cochin Hand Functional Scale (CHFS), Short-Form 36 Health Survey (SF-36); Scleroderma Health Assessment Questionnaire Disability Index (SHAQ-DI); lung function; lung ultrasound; handgrip; Glittre Activities of Daily Living test. Thus, it is expected that patients with SS will benefit significantly, with a consequent improvement in musculoskeletal function and , functional capacity and health-related quality of life.

DETAILED DESCRIPTION:
In the current epidemiological context, chronic diseases affect very specific and neglected populations. In addition to their rarity, these diseases are characterized by a progressive increase in the life expectancy of their patients and important functional limitations due to their multisystemic character. In this context, there is Systemic Sclerosis - SSc (or Scleroderma), which presents peculiar clinical and functional aspects that limit the activities of daily living (ADL) of patients. Although the focus of SSc treatment is the clinical control of the disease, a new perspective must be given to the aspect of functional rehabilitation. Therefore, this study proposes a therapist-oriented home rehabilitation program (TOHR) for these patients. Considering that in SSc the hands are predominantly affected, and that functional incapacity of the hands is the main component of global incapacity in this population, the ADL-Glittre test has been used as a submaximal functional capacity test as it involves lower and upper limbs, as well as diversified tasks, coming closer to the activities that the individual does in its usual environment. Thus, the present study aims to evaluate the effects of a TOHR program on the functional capacity of patients with SSc, through the ADL-Glittre test, considering the impact of hand function, peripheral muscle strength, pulmonary function and quality of life. For this, women with SSc will be evaluated, submitted to the following tests: Cochin Hand Functional Scale, Short-Form 36 Health Survey; Scleroderma Health Assessment Questionnaire Disability Index; handgrip dynamometry; impulse oscillometry technique; spirometry; lung ultrasound and ADL-Glittre test. Additionally, patients will undergo a 12-week TOHR protocol. At the end of this period, all evaluations will be repeated. This will be a prospective, longitudinal study, with quantitative assessment of sample data. The aim of the study is to support the applicability of a TOHR program in women with SSc.

ELIGIBILITY:
Inclusion Criteria:

* Women with Scleroderma, older than 18 years
* Clinical stability
* Signature of the Informed Consent Term (TCLE)

Exclusion Criteria:

* Patients with inability to perform the Glittre Activities of Daily Living test
* Patients who have cognitive impairment by mini mental state examination (MEEN).
* Abandonment of treatment of scleroderma during the application of the protocol.
* Uncontrolled hypertension (> 180/100 mmHg with medication use)
* Use of psychotropic drugs
* Any significant limitations due to osteoarthropathy
* History of surgery in the previous six months with exercise restriction
* IPAQ with very active classification

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Scleroderma is more frequent in females than in males.
Enrollment: 104 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional capacity through the Glittre Activities of Daily Living test (ADL-Glittre test) before and after the execution of the treatment plan | twelve weeks
  Performed as proposed by Skumlien et al. (2006), the participant must complete 5 laps in the shortest possible time. The test consists of carrying a backpack containing a 2.5 kg weight completing a circuit with the following activities. The participant rises from a seated position and walks on a 10-m flat course, interposed halfway by a stairway with 2 steps to ascend and 2 to descend. After completing the course, the individual approaches a 2-teir shelf containing 3 objects weighing 1 kg each, placed on the highest shelf (shoulder height), that must be moved 1 by 1 to the bottom shelf (waist height) and then down to the floor. Then, the objects are placed on the bottom shelf again and finally on the top shelf. Then, the individual turns and walks back over the course; immediately after completion of 1 lap, another lap is started, completing the same circuit. The instructions are standardized, and there is no incentive during the test. Two tests are performed with a minim.

SECONDARY OUTCOMES:
Peripheral muscle function before and after the execution of the treatment plan | twelve weeks
  Isometric handgrip strength (IHGS) was measured using a hydraulic isometric dynamometer (SH5001, Saehan Corporation, Korea) with the hand on the dominant side of the body. Participants were comfortably seated in a chair with no arm rest, with the feet flat on the floor and hips and knees flexed at 90°. The shoulder was adducted, the elbow was flexed at 90º, and the forearm was in a neutral position; the wrist position could vary between 0-30º of extension and 0-15º of ulnar deviation. The participants were then instructed to perform 3 maximum voluntary contractions with a 60-s interval in between. The tests followed the standards established by the American Society of Hand Therapists. The highest recorded value among the 3 measurements was considered.
Cochin Hand Functional Scale (CHFS) | twelve weeks
  The CHFS was used to assess the level of hand ability and functionality in the performance of daily activities. The CHFS contains 18 items concerning ADLs that require manual skills, such as cooking, dressing and personal hygiene. This scale takes approximately 3 min to complete and considers only the experiences of the individual during the past month. Each item has 6 possible answers, as follows: without difficulty (0); with very little difficulty (1); with some difficulty (2); with much difficulty (3); nearly impossible to do (4); and impossible to do (5). The score is the sum of all items and ranges from 0 to 90; the higher the score is, the greater the hand dysfunction.
Quality of life related to activities of daily living through the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) before and after the execution of the treatment plan. | twelve weeks
  The 36-Item Short Form Survey (SF-36) is an oft-used, well-researched, self-reported measure of health. It stems from a study called the Medical Outcomes Study. Patients or individuals are asked to fill out the questionnaire (tick boxes) by themselves and then it is scored by a researcher. It contains the 36 questions and answers in the bodily pain and general health domains.Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high QOL. Two component scores can also be tallied; a physical component summary and a mental component summary.
Pulmonary Function Tests before and after the execution of the treatment plan | twelve weeks
  Impulse oscillometry (IOS) will use an impulse oscillometer (Quark i2m, Cosmed, Rome, Italy). IOS measures the respiratory system impedance (Zrs) composed of the respiratory system resistance and the respiratory system reactance. The minimum acceptable coherence values will be those ≥ 0.9 Hz. (RIBEIRO et al, 2018) Participants will also perform spirometry (VT 130 SL, Codax Ltda, Rio de Janeiro, Brazil), using standardization made by the American Thoracic Society/European Respiratory Society. The predicted values of FVC, expiratory volume in one second (FEV1) and forced expiratory flow between 25-75% of FVC (FEF25-75%) will be calculated according to the equations of Pereira et al (2007) and the results will be expressed as percentages of the predicted values. Obstructive disorder will be defined by an FEV1/FVC ratio <70%, while a restrictive disorder will be inferred by a FVC <80% predicted in the absence of reduced expiratory flows.
Lung ultrassound before and after the execution of the treatment plan | twelve weeks
  Using an Aplio XG Aplio XG equipment (Toshiba Medical Systems, Tokyo, Japan), with a 7.5-10 MHz multifrequency linear transducer or a 3.5-5 MHz convex transducer in B mode, the USP exams will be performed on the same day as the TFP. Following a 12-zone protocol and with participants in a seated position, the USP exams will be performed in 6 areas of each hemithorax (two anterior, two lateral and two posterior). USP images will be examined for the evaluation of the following signs: B lines > 2, coalescent B lines and subpleural consolidations. In order to classify the lung injury, in each of these 6 areas, weights ranging from 1 to 3 will be assigned for each finding in the USP, as follows: 1 = lines B > 2; 2 = coalescent B lines; and 3 = subpleural consolidations). The sum of all 6 areas evaluated at USP will represent the aeration score, which may vary between 0-18 points. (SOUMMER et al., 2012; TUNG-CHEN et al., 2020)
Disability assessment using the Scleroderma Health Assessment Questionnaire Disability Index (SHAQ-DI) before and after the execution of the treatment plan | twelve weeks
  The SHAQ-DI will be used to assess the participants' level of physical function. This questionnaire includes questions related to fine movements of the upper extremities and motor activities of the lower limbs (BRUCE & FRIES, 2003). There are 20 questions divided into 8 categories that represent a comprehensive set of functional activities performed in the last 7 days, including the ability to dress, stand up, eat, walk, perform personal hygiene, reach or grab something, and perform usual activities . To quantify the values found, the SHAQ-DI has a 26 score ranging from 0 (no disability) to 3 (maximum disability). The total score is the average of the scores of the 8 categories.

CONTACTS AND LOCATIONS:
Locations (1):
- Centro Universitário Augusto Motta, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhajeri H, Hudson M, Fritzler M, Pope J, Tatibouet S, Markland J, Robinson D, Jones N, Khalidi N, Docherty P, Kaminska E, Masetto A, Sutton E, Mathieu JP, Ligier S, Grodzicky T, LeClercq S, Thorne C, Gyger G, Smith D, Fortin PR, Larche M, Baron M. 2013 American College of Rheumatology/European League against rheumatism classification criteria for systemic sclerosis outperform the 1980 criteria: data from the Canadian Scleroderma Research Group. Arthritis Care Res (Hoboken). 2015 Apr;67(4):582-7. doi: 10.1002/acr.22451. PMID 25233870
- [Background] Avouac J, Walker U, Tyndall A, Kahan A, Matucci-Cerinic M, Allanore Y; EUSTAR; Miniati I, Muller A, Iannone F, Distler O, Becvar R, Sierakowsky S, Kowal-Bielecka O, Coelho P, Cabane J, Cutolo M, Shoenfeld Y, Valentini G, Rovensky J, Riemekasten G, Vlachoyiannopoulos P, Caporali R, Jiri S, Inanc M, Zimmermann Gorska I, Carreira P, Novak S, Czirjak L, Oliveira Ramos F, Jendro M, Chizzolini C, Kucharz EJ, Richter J, Cozzi F, Rozman B, Mallia CM, Gabrielli A, Farge D, Kiener HP, Schoffel D, Airo P, Wollheim F, Martinovic D, Trotta F, Jablonska S, Reich K, Bombardieri S, Siakka P, Pellerito R, Bambara LM, Morovic-Vergles J, Denton C, Hinrichs R, Van den Hoogen F, Damjanov N, Kotter I, Ortiz V, Heitmann S, Krasowska D, Seidel M, Hasler P, Van Laar JM, Kaltwasser JP, Foeldvari I, Juan Mas A, Bajocchi G, Wislowska M, Pereira Da Silva JA, Jacobsen S, Worm M, Graniger W, Kuhn A, Stankovic A, Cossutta R, Majdan M, Damjanovska Rajcevska L, Tikly M, Nasonov EL, Steinbrink K, Herrick A, Muller-Ladner U, Dinc A, Scorza R, Sondergaard K, Indiveri F, Nielsen H, Szekanecz Z, Silver RM, Antivalle M, Espinosa IB, Garcia de la Pena Lefebvre P, Midtvedt O, Launay D, Valesini F, Tuvik P, Ionescu RM, Del Papa N, Pinto S, Wigley F, Mihai C, Sinziana Capranu M, Sunderkotter C, Jun JB, Alhasani S, Distler JH, Ton E, Soukup T, Seibold J, Zeni S, Nash P, Mouthon L, De Keyser F, Duruoz MT, Cantatore FP, Strauss G, von Mulhen CA, Pozzi MR, Eyerich K, Szechinski J, Keiserman M, Houssiau FA, Roman-Ivorra JA, Krummel-Lorenz B, Aringer M, Westhovens R, Bellisai F, Mayer M, Stoeckl F, Uprus M, Volpe A, Buslau M, Yavuz S, Granel B, Valderilio Feijo A, Del Galdo F, Popa S, Zenone T, Ricardo Machado X, Pileckyte M, Stebbings S, Mathieu A, Tulli A, Tourinho T, Souza R, Acayaba de Toledo R, Stamp L, Solanki K, Veale D, Francisco Marques Neto J, Bagnato GF, Loyo E, Toloza S, Li M, Ahmed Abdel Atty Mohamed W, Cobankara V, Olas J, Salsano F, Oksel F, Tanaseanu CM, Foti R, Ancuta C, Vonk M, Caramashi P, Beretta L, Balbir A, Chiala A, Pasalic Simic K, Ghio M, Stamenkovic B, Rednic S, Host N, Pellerito R, Hachulla E, Furst DE. Characteristics of joint involvement and relationships with systemic inflammation in systemic sclerosis: results from the EULAR Scleroderma Trial and Research Group (EUSTAR) database. J Rheumatol. 2010 Jul;37(7):1488-501. doi: 10.3899/jrheum.091165. Epub 2010 Jun 15. PMID 20551097
- [Background] Barsotti S, Stagnaro C, d'Ascanio A, Della Rossa A. One year in review 2016: systemic sclerosis. Clin Exp Rheumatol. 2016 Sep-Oct;34 Suppl 100(5):3-13. Epub 2016 Jul 18. PMID 27463613
- [Background] Bellando-Randone S, Matucci-Cerinic M. Very Early Systemic Sclerosis and Pre-systemic Sclerosis: Definition, Recognition, Clinical Relevance and Future Directions. Curr Rheumatol Rep. 2017 Sep 18;19(10):65. doi: 10.1007/s11926-017-0684-2. PMID 28921059
- [Background] Boutou AK, Pitsiou GG, Siakka P, Dimitroulas T, Paspala A, Sourla E, Chavouzis N, Garyfallos A, Argyropoulou P, Stanopoulos I. Phenotyping Exercise Limitation in Systemic Sclerosis: The Use of Cardiopulmonary Exercise Testing. Respiration. 2016;91(2):115-23. doi: 10.1159/000442888. Epub 2016 Jan 6. PMID 26731293
- [Background] Brower LM, Poole JL. Reliability and validity of the Duruoz Hand Index in persons with systemic sclerosis (scleroderma). Arthritis Rheum. 2004 Oct 15;51(5):805-9. doi: 10.1002/art.20701. PMID 15478150
- [Background] Bruce B, Fries JF. The Stanford Health Assessment Questionnaire: dimensions and practical applications. Health Qual Life Outcomes. 2003 Jun 9;1:20. doi: 10.1186/1477-7525-1-20. PMID 12831398
- [Background] Cella DF, Bonomi AE. Measuring quality of life: 1995 update. Oncology (Williston Park). 1995 Nov;9(11 Suppl):47-60. PMID 8608056
- [Background] Coulter CL, Scarvell JM, Neeman TM, Smith PN. Physiotherapist-directed rehabilitation exercises in the outpatient or home setting improve strength, gait speed and cadence after elective total hip replacement: a systematic review. J Physiother. 2013 Dec;59(4):219-26. doi: 10.1016/S1836-9553(13)70198-X. PMID 24287215
- [Background] Crosby CA, Wehbe MA, Mawr B. Hand strength: normative values. J Hand Surg Am. 1994 Jul;19(4):665-70. doi: 10.1016/0363-5023(94)90280-1. PMID 7963331
- [Background] de Oliveira NC, Portes LA, Pettersson H, Alexanderson H, Bostrom C. Aerobic and resistance exercise in systemic sclerosis: State of the art. Musculoskeletal Care. 2017 Dec;15(4):316-323. doi: 10.1002/msc.1185. Epub 2017 Apr 5. PMID 28378937
- [Background] Dechman G, Scherer SA. Outcome Measures in Cardiopulmonary Physical Therapy: Focus on the Glittre ADL-Test for People with Chronic Obstructive Pulmonary Disease. Cardiopulm Phys Ther J. 2008 Dec;19(4):115-8. No abstract available. PMID 20467508
- [Background] Duruoz MT, Poiraudeau S, Fermanian J, Menkes CJ, Amor B, Dougados M, Revel M. Development and validation of a rheumatoid hand functional disability scale that assesses functional handicap. J Rheumatol. 1996 Jul;23(7):1167-72. PMID 8823687
- [Background] Fernandes-Andrade AA, Britto RR, Soares DCM, Velloso M, Pereira DAG. Evaluation of the Glittre-ADL test as an instrument for classifying functional capacity of individuals with cardiovascular diseases. Braz J Phys Ther. 2017 Sep-Oct;21(5):321-328. doi: 10.1016/j.bjpt.2017.06.001. Epub 2017 Jul 3. PMID 28711380
- [Background] Ganderton L, Jenkins S, Gain K, Fowler R, Winship P, Lunt D, Gabbay E. Short term effects of exercise training on exercise capacity and quality of life in patients with pulmonary arterial hypertension: protocol for a randomised controlled trial. BMC Pulm Med. 2011 May 23;11:25. doi: 10.1186/1471-2466-11-25. PMID 21600062
- [Background] Ingegnoli F, Boracchi P, Ambrogi F, Gualtierotti R, Galbiati V, Meroni PL. Hand impairment in systemic sclerosis: association of different hand indices with organ involvement. Scand J Rheumatol. 2010;39(5):393-7. doi: 10.3109/03009741003629028. PMID 20476855
- [Background] Justo AC, Guimaraes FS, Ferreira AS, Soares MS, Bunn PS, Lopes AJ. Muscle function in women with systemic sclerosis: Association with fatigue and general physical function. Clin Biomech (Bristol). 2017 Aug;47:33-39. doi: 10.1016/j.clinbiomech.2017.05.011. Epub 2017 May 26. PMID 28575704
- [Background] Khanna D, Kowal-Bielecka O, Khanna PP, Lapinska A, Asch SM, Wenger N, Brown KK, Clements PJ, Getzug T, Mayes MD, Medsger TA, Oudiz R, Simms R, Steen V, Maranian P, Furst DE. Quality indicator set for systemic sclerosis. Clin Exp Rheumatol. 2011 Mar-Apr;29(2 Suppl 65):S33-9. Epub 2011 May 16. PMID 21586216
- [Background] Lima TRL, Kasuki L, Gadelha M, Lopes AJ. Physical exercise improves functional capacity and quality of life in patients with acromegaly: a 12-week follow-up study. Endocrine. 2019 Nov;66(2):301-309. doi: 10.1007/s12020-019-02011-x. Epub 2019 Jul 17. PMID 31317523
- [Background] Gasho CJ, Torralba KD, Chooljian DM, Cohen A, Dinh VA. Impact of a lung ultrasound course for rheumatology specialists (IMPACT-2). Clin Exp Rheumatol. 2019 May-Jun;37(3):380-384. Epub 2018 Aug 29. PMID 30183605
- [Background] Wang Y, Gargani L, Barskova T, Furst DE, Cerinic MM. Usefulness of lung ultrasound B-lines in connective tissue disease-associated interstitial lung disease: a literature review. Arthritis Res Ther. 2017 Sep 18;19(1):206. doi: 10.1186/s13075-017-1409-7. PMID 28923086
- [Background] Landim SF, Bertolo MB, Marcatto de Abreu MF, Del Rio AP, Mazon CC, Marques-Neto JF, Poole JL, de Paiva Magalhaes E. The evaluation of a home-based program for hands in patients with systemic sclerosis. J Hand Ther. 2019 Jul-Sep;32(3):313-321. doi: 10.1016/j.jht.2017.10.013. Epub 2017 Dec 1. PMID 29198478
- [Background] Levis AW, Harel D, Kwakkenbos L, Carrier ME, Mouthon L, Poiraudeau S, Bartlett SJ, Khanna D, Malcarne VL, Sauve M, van den Ende CH, Poole JL, Schouffoer AA, Welling J, Thombs BD; the Scleroderma Patient-Centered Intervention Network Investigators. Using Optimal Test Assembly Methods for Shortening Patient-Reported Outcome Measures: Development and Validation of the Cochin Hand Function Scale-6: A Scleroderma Patient-Centered Intervention Network Cohort Study. Arthritis Care Res (Hoboken). 2016 Nov;68(11):1704-1713. doi: 10.1002/acr.22893. Epub 2016 Oct 9. PMID 27015290
- [Background] Li L, Cui Y, Chen S, Zhao Q, Fu T, Ji J, Li L, Gu Z. The impact of systemic sclerosis on health-related quality of life assessed by SF-36: A systematic review and meta-analysis. Int J Rheum Dis. 2018 Nov;21(11):1884-1893. doi: 10.1111/1756-185X.13438. Epub 2018 Nov 14. PMID 30428506
- [Background] Lima TR, Guimaraes FS, Carvalho MN, Sousa TL, Menezes SL, Lopes AJ. Lower limb muscle strength is associated with functional performance and quality of life in patients with systemic sclerosis. Braz J Phys Ther. 2015 Mar-Apr;19(2):129-36. doi: 10.1590/bjpt-rbf.2014.0084. Epub 2015 Mar 13. PMID 25789555
- [Background] Lopes AJ, Capone D, Mogami R, Menezes SL, Guimaraes FS, Levy RA. Systemic sclerosis-associated interstitial pneumonia: evaluation of pulmonary function over a five-year period. J Bras Pneumol. 2011 Mar-Apr;37(2):144-51. doi: 10.1590/s1806-37132011000200003. English, Portuguese. PMID 21537649
- [Background] Lopes AJ, Justo AC, Ferreira AS, Guimaraes FS. Systemic sclerosis: Association between physical function, handgrip strength and pulmonary function. J Bodyw Mov Ther. 2017 Oct;21(4):972-977. doi: 10.1016/j.jbmt.2017.03.018. Epub 2017 Mar 29. PMID 29037654
- [Background] Maddali-Bongi S, Del Rosso A. Systemic sclerosis: rehabilitation as a tool to cope with disability. Clin Exp Rheumatol. 2016 Sep-Oct;34 Suppl 100(5):162-169. Epub 2016 Jul 4. PMID 27384349
- [Background] Mitropoulos A, Gumber A, Crank H, Akil M, Klonizakis M. The effects of upper and lower limb exercise on the microvascular reactivity in limited cutaneous systemic sclerosis patients. Arthritis Res Ther. 2018 Jun 5;20(1):112. doi: 10.1186/s13075-018-1605-0. PMID 29871697
- [Background] Morrisroe KB, Nikpour M, Proudman SM. Musculoskeletal Manifestations of Systemic Sclerosis. Rheum Dis Clin North Am. 2015 Aug;41(3):507-18. doi: 10.1016/j.rdc.2015.04.011. Epub 2015 May 26. PMID 26210132
- [Background] Morrisroe K, Stevens W, Huq M, Prior D, Sahhar J, Ngian GS, Celermajer D, Zochling J, Proudman S, Nikpour M; Australian Scleroderma Interest Group (ASIG). Survival and quality of life in incident systemic sclerosis-related pulmonary arterial hypertension. Arthritis Res Ther. 2017 Jun 2;19(1):122. doi: 10.1186/s13075-017-1341-x. PMID 28576149
- [Background] Mouthon L, Mestre-Stanislas C, Berezne A, Rannou F, Guilpain P, Revel M, Pagnoux C, Guillevin L, Fermanian J, Poiraudeau S. Impact of digital ulcers on disability and health-related quality of life in systemic sclerosis. Ann Rheum Dis. 2010 Jan;69(1):214-7. doi: 10.1136/ard.2008.094193. PMID 19221115
- [Background] Murphy SL, Barber MW, Homer K, Dodge C, Cutter GR, Khanna D. Occupational Therapy Treatment to Improve Upper Extremity Function in Individuals with Early Systemic Sclerosis: A Pilot Study. Arthritis Care Res (Hoboken). 2018 Nov;70(11):1653-1660. doi: 10.1002/acr.23522. PMID 29381834
- [Background] Paik JJ, Wigley FM, Mejia AF, Hummers LK. Independent Association of Severity of Muscle Weakness With Disability as Measured by the Health Assessment Questionnaire Disability Index in Scleroderma. Arthritis Care Res (Hoboken). 2016 Nov;68(11):1695-1703. doi: 10.1002/acr.22870. Epub 2016 Oct 9. PMID 26881982
- [Background] Peytrignet S, Denton CP, Lunt M, Hesselstrand R, Mouthon L, Silman A, Pan X, Brown E, Czirjak L, Distler JHW, Distler O, Fligelstone K, Gregory WJ, Ochiel R, Vonk M, Ancuta C, Ong VH, Farge D, Hudson M, Matucci-Cerinic M, Balbir-Gurman A, Midtvedt O, Jordan AC, Stevens W, Moinzadeh P, Hall FC, Agard C, Anderson ME, Diot E, Madhok R, Akil M, Buch MH, Chung L, Damjanov N, Gunawardena H, Lanyon P, Ahmad Y, Chakravarty K, Jacobsen S, MacGregor AJ, McHugh N, Muller-Ladner U, Riemekasten G, Becker M, Roddy J, Carreira PE, Fauchais AL, Hachulla E, Hamilton J, Inanc M, McLaren JS, van Laar JM, Pathare S, Proudman S, Rudin A, Sahhar J, Coppere B, Serratrice C, Sheeran T, Veale DJ, Grange C, Trad GS, Herrick AL. Disability, fatigue, pain and their associates in early diffuse cutaneous systemic sclerosis: the European Scleroderma Observational Study. Rheumatology (Oxford). 2018 Feb 1;57(2):370-381. doi: 10.1093/rheumatology/kex410. PMID 29207002
- [Background] Racine M, Hudson M, Baron M, Nielson WR; Canadian Scleroderma Research Group. The Impact of Pain and Itch on Functioning and Health-Related Quality of Life in Systemic Sclerosis: An Exploratory Study. J Pain Symptom Manage. 2016 Jul;52(1):43-53. doi: 10.1016/j.jpainsymman.2015.12.314. Epub 2016 Feb 11. PMID 26876159
- [Background] Rannou F, Poiraudeau S, Berezne A, Baubet T, Le-Guern V, Cabane J, Guillevin L, Revel M, Fermanian J, Mouthon L. Assessing disability and quality of life in systemic sclerosis: construct validities of the Cochin Hand Function Scale, Health Assessment Questionnaire (HAQ), Systemic Sclerosis HAQ, and Medical Outcomes Study 36-Item Short Form Health Survey. Arthritis Rheum. 2007 Feb 15;57(1):94-102. doi: 10.1002/art.22468. PMID 17266096
- [Background] Ranque B, Authier FJ, Berezne A, Guillevin L, Mouthon L. Systemic sclerosis-associated myopathy. Ann N Y Acad Sci. 2007 Jun;1108:268-82. doi: 10.1196/annals.1422.029. PMID 17899625
- [Background] Ranque B, Authier FJ, Le-Guern V, Pagnoux C, Berezne A, Allanore Y, Launay D, Hachulla E, Kahan A, Cabane J, Gherardi R, Guillevin L, Mouthon L. A descriptive and prognostic study of systemic sclerosis-associated myopathies. Ann Rheum Dis. 2009 Sep;68(9):1474-7. doi: 10.1136/ard.2008.095919. Epub 2008 Dec 3. PMID 19054827
- [Background] Reis CMD, Karloh M, Fonseca FR, Biscaro RRM, Mazo GZ, Mayer AF. Functional capacity measurement: reference equations for the Glittre Activities of Daily Living test. J Bras Pneumol. 2018 Sep-Oct;44(5):370-377. doi: 10.1590/S1806-37562017000000118. Epub 2018 Jul 16. PMID 30020345
- [Background] Salaffi F, Di Carlo M, Carotti M, Farah S, Ciapetti A, Gutierrez M. The impact of different rheumatic diseases on health-related quality of life: a comparison with a selected sample of healthy individuals using SF-36 questionnaire, EQ-5D and SF-6D utility values. Acta Biomed. 2019 Jan 15;89(4):541-557. doi: 10.23750/abm.v89i4.7298. PMID 30657123
- [Background] Sandqvist G, Eklund M, Akesson A, Nordenskiold U. Daily activities and hand function in women with scleroderma. Scand J Rheumatol. 2004;33(2):102-7. doi: 10.1080/03009740410006060. PMID 15163111
- [Background] Schorpion A, Shenin M, Neubauer R, Derk CT. A prospective, open-label, non-comparative study of ambrisentan with anti-fibrotic agent combination therapy in the treatment of diffuse systemic sclerosis. BMC Rheumatol. 2018 May 15;2:13. doi: 10.1186/s41927-018-0021-z. eCollection 2018. PMID 30886964
- [Background] Skumlien S, Hagelund T, Bjortuft O, Ryg MS. A field test of functional status as performance of activities of daily living in COPD patients. Respir Med. 2006 Feb;100(2):316-23. doi: 10.1016/j.rmed.2005.04.022. Epub 2005 Jun 6. PMID 15941658
- [Background] Sultan N, Pope JE, Clements PJ; Scleroderma Trials Study Group. The health assessment questionnaire (HAQ) is strongly predictive of good outcome in early diffuse scleroderma: results from an analysis of two randomized controlled trials in early diffuse scleroderma. Rheumatology (Oxford). 2004 Apr;43(4):472-8. doi: 10.1093/rheumatology/keh070. Epub 2003 Dec 16. PMID 14679295
- [Background] van den Hoogen F, Khanna D, Fransen J, Johnson SR, Baron M, Tyndall A, Matucci-Cerinic M, Naden RP, Medsger TA Jr, Carreira PE, Riemekasten G, Clements PJ, Denton CP, Distler O, Allanore Y, Furst DE, Gabrielli A, Mayes MD, van Laar JM, Seibold JR, Czirjak L, Steen VD, Inanc M, Kowal-Bielecka O, Muller-Ladner U, Valentini G, Veale DJ, Vonk MC, Walker UA, Chung L, Collier DH, Ellen Csuka M, Fessler BJ, Guiducci S, Herrick A, Hsu VM, Jimenez S, Kahaleh B, Merkel PA, Sierakowski S, Silver RM, Simms RW, Varga J, Pope JE. 2013 classification criteria for systemic sclerosis: an American college of rheumatology/European league against rheumatism collaborative initiative. Ann Rheum Dis. 2013 Nov;72(11):1747-55. doi: 10.1136/annrheumdis-2013-204424. PMID 24092682
- [Background] Varga J, Hinchcliff M. Connective tissue diseases: systemic sclerosis: beyond limited and diffuse subsets? Nat Rev Rheumatol. 2014 Apr;10(4):200-2. doi: 10.1038/nrrheum.2014.22. Epub 2014 Feb 18. PMID 24535544
- [Background] Walker UA, Tyndall A, Czirjak L, Denton C, Farge-Bancel D, Kowal-Bielecka O, Muller-Ladner U, Bocelli-Tyndall C, Matucci-Cerinic M. Clinical risk assessment of organ manifestations in systemic sclerosis: a report from the EULAR Scleroderma Trials And Research group database. Ann Rheum Dis. 2007 Jun;66(6):754-63. doi: 10.1136/ard.2006.062901. Epub 2007 Jan 18. PMID 17234652
- [Background] Wollheim FA. Classification of systemic sclerosis. Visions and reality. Rheumatology (Oxford). 2005 Oct;44(10):1212-6. doi: 10.1093/rheumatology/keh671. Epub 2005 May 3. PMID 15870151
- [Derived] de Alegria SG, Litrento PF, de Oliveira Farias I, Mafort TT, Lopes AJ. Can home rehabilitation impact impulse oscillometry and lung ultrasound findings in patients with scleroderma-associated interstitial lung disease? A pilot study. BMC Res Notes. 2022 May 15;15(1):176. doi: 10.1186/s13104-022-06064-6. PMID 35570301
- See also: Translation, cultural adaptation and reproducibility of the Cochin Hand Functional Scale questionnaire for Brazil — https://doi.org/10.1590/S1807-59322011000500004
- See also: Pereira CAC. Espirometria. J Bras Pneumol. 2002; 28(Supl. 3): 1-82. — https://www.google.com/url?sa=t&rct=j&q=&esrc=s&source=web&cd=&cad=rja&uact=8&ved=2ahUKEwiYpu-H8tPwAhW-qJUCHRUjANgQFjAAegQIAhAD&url=http%3A%2F%2Fwww.saude.ufpr.br%2Fportal%2Flabsim%2Fwp-content%2Fuploads%2Fsites%2F23%2F2016%2F07%2FSuple_139_45_11-Espirometria.pdf&usg=AOvVaw1UGXp51DUZsTOXA2rjdVOy